CLINICAL TRIAL: NCT07085026
Title: The Effect of Yoga Practiced in the Third Trimester on Sleep and Stress
Brief Title: Effects of Yoga on Sleep and Stress in the Third Trimester of Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gözde Şengün, Master's Degree Student with Thesis, Istanbul University- Cerrahpasa Midwifery Department, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IUC-SBF-GŞ-01
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Stress
Keywords: yoga; sleep; stress; pregnancy; third trimester

STUDY DESIGN:
Intervention Model Description: Pregnant participants will be randomly assigned to two groups in a 1:1 ratio. The intervention group will receive a yoga program in accordance with the WHO guideline recommendations, while the control group will receive no intervention and will continue with routine care.
Masking Description: Because of the behavioral and observable characteristics of the intervention (yoga in the third trimester of pregnancy), neither assessment nor blinding of investigators was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will practice yoga in accordance with the WHO guideline recommendations.
  Interventions: Behavioral: Yoga Intervention
- Control Group (No Intervention): Participants in this group will not receive yoga; routine care will be provided.

INTERVENTIONS:
Behavioral: Yoga Intervention — There are studies that have evaluated the effects of prenatal yoga on sleep. None of these studies have reported any negative effects of yoga on pregnancy. In all studies, yoga practice was applied with varying frequencies, durations, and techniques. However, no research has been found that evaluates the effects of a yoga program conducted in accordance with the World Health Organization (WHO) guideline recommendations on both sleep and stress. Therefore, the aim of this study is to evaluate the effects of yoga, practiced during the third trimester of pregnancy in line with WHO guideline recommendations, on sleep and stress.
  Arms: Intervention Group

SUMMARY:
Many physiological and psychological changes occur during pregnancy. Sleep and stress are among these changes and can negatively impact the pregnancy process. Yoga can improve sleep quality and stress levels during pregnancy. The purpose of this study was to evaluate the effects of yoga, implemented in the third trimester of pregnancy according to World Health Organization guidelines, on sleep and stress.

DETAILED DESCRIPTION:
Pregnancy is defined as a period of both physiological and psychological changes in women. Although pregnancy and childbirth are natural processes, the physical, mental, and emotional adaptive changes that occur during this time can significantly impact a woman's health and pregnancy outcomes. Sleep problems are common during pregnancy. Toward the end of pregnancy, women often experience frequent nighttime awakenings, insomnia, and restless sleep. During pregnancy, women undergo bio-physio-psychosocial changes that can lead to increased stress. In order to prevent adverse outcomes, it is important to manage stress in pregnant women and implement interventions aimed at reducing high cortisol levels.

Yoga can be defined as a system of stretching exercises and postures (asanas) combined with deep breathing (pranayama) and meditation, aiming to unify the mind, body, and spirit.

There are studies that have evaluated the effects of yoga practice during pregnancy on sleep and stress. None of these studies have reported any negative effects of yoga on pregnancy. In all studies, yoga was applied with varying frequencies, durations, and techniques. However, no study has been found that evaluates the effects of a yoga program conducted in accordance with the recommendations of the World Health Organization (WHO, 2023) on both sleep and stress. Therefore, the aim of this study is to evaluate the effects of yoga, implemented during the third trimester of pregnancy in line with WHO guideline recommendations, on sleep and stress.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreed to participate in the study,
* Aged between 18 and 35 years,
* In the third trimester of pregnancy (between 29 and 42 weeks of gestation),
* Able to read and write in Turkish,
* No prior experience with yoga practice.

Exclusion Criteria:

* High-risk pregnancy,
* In the first or second trimester,
* Multiple pregnancy,
* Any condition that prevents yoga practice (e.g., restrictions on physical activity),
* Previous experience with yoga practice

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | It will be assessed at baseline (in the third trimester of pregnancy) and on day 30 after the yoga intervention.
  Sleep quality is measured by the Pittsburgh Sleep Quality Index (PSQI).
  The Pittsburgh Sleep Quality Index (PSQI) was developed to assess sleep quality and sleep disturbances over the past month. It consists of a total of 24 questions, 19 of which are self-rated items. The remaining 5 questions are used for clinical evaluation and are not included in the scoring. Each item in the scale is rated on a scale from 0 to 3. From the 19 self-rated items, 7 component scores are derived. Some components are based on a single item, while others are formed by combining several items. These components are: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The total score of the scale is obtained by summing the scores of these 7 components. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A total score greater than 5 indicates "poor sleep quality."

SECONDARY OUTCOMES:
Perceived Stress Level | It will be assessed at baseline (in the third trimester of pregnancy) and on day 30 after the yoga intervention.
  Maternal stress level assessed using the Perceived Stress Scale (PSS).
  The Perceived Stress Scale (PSS) was developed to assess perceived stress over the past month. It consists of 14 items and is rated on a 5-point Likert scale ranging from "Never (0)" to "Very Often (4)". Seven of the items, which are positively stated, are reverse scored. The total score of the PSS-14 ranges from 0 to 56, with higher scores indicating greater levels of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay TÜLAY Yılmaz, Associate Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine Prof. Dr. Murat Dilmener Hospital, Istanbul, Bakirköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No